CLINICAL TRIAL: NCT02793271
Title: Reducing Stigma Among Healthcare Providers to Improve Mental Health Services: RESHAPE-mh Protocol for a Feasibility and Acceptability Pilot Cluster Randomized Control Trial
Brief Title: Reducing Stigma Among Healthcare Providers to Improve Mental Health Services
Acronym: RESHAPE-mh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandon A Kohrt, MD, PhD (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Brandon A Kohrt, MD, PhD, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00055042; K01MH104310 (NIH)
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Mental Disorders
Keywords: Depression; Primary Health Care; Social Stigma; Stereotyping; Health Care Quality; Access; Evaluation
MeSH Terms: conditions — Mental Disorders; Depression; Social Stigma; Stereotyping | interventions — PRIME protocol; Mental Health Services; Primary Health Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRIME (Active Comparator): The behavioral intervention will be the PRIME/mhGAP training. This is standard mental health training for prescribers (primary care workers who can prescribe psychotropic medication, e.g., health assistants) and non-prescribers (primary care workers who cannot prescribe medications, e.g., auxilliary nurse midwives). For prescribers, training includes introduction to psychosocial techniques and mhGAP. For non-prescribers, training includes psychosocial techniques.
  Interventions: Behavioral: PRIME/mhGAP
- PRIME+RESHAPE (Experimental): The behavioral intervention will be the PRIME/mhGAP training plus the RESHAPE training adjunct. This is the PRIME training plus social contact component in which mental health service users participate as training co-facilitators. The intended goal of the additional component is to reduce stigma against persons with mental illness.
  Interventions: Behavioral: RESHAPE; Behavioral: PRIME/mhGAP

INTERVENTIONS:
Behavioral: RESHAPE — Mental health services users and primary care workers who have previously completed the training are trained using PhotoVoice and other techniques to participate as co-facilitators. They participate in introductions to the intervention, myth busting, recovery stories, psychosocial communication role plays, and collaborative activities addressing challenges and barriers to task sharing/ task shifting mental health services in primary care.
  Other Names: Social contact anti-stigma behavioral intervention
  Arms: PRIME+RESHAPE
Behavioral: PRIME/mhGAP — Primary care workers are trained using the mental health Global Action Programme (mhGAP) to identify and treat mental disorders in primary care. Primary care "prescribers" (those who can administer psychotropic medication) are trained to treat disorders including depression, alcohol use disorder, psychosis / schizophrenia, and epilepsy. "Non-prescribers" (primary care workers not authorized to dispense medications) are trained to deliver psychosocial and psychological interventions.
  Other Names: Mental health services for primary care

SUMMARY:
A growing number of trials have demonstrated treatment effectiveness for people with mental illness (PWMI) by non-specialist providers, such as primary care and community health workers, in low-resource settings. A barrier to scaling up these evidence-based practices is the limited uptake from trainings into service provision and lack of fidelity to evidence-based practices among non-specialists. This arises, in part, from stigma among non-specialists against PWMI. Therefore, interventions are needed to address attitudes among non-specialists. To address this gap, REducing Stigma among HeAlthcare Providers to improvE Mental Health services (RESHAPE-mh), is an intervention for non-specialists in which social contact with PWMI is added to training and supervision programs. A pilot cluster randomized control trial will address primary objectives including trainees' perspectives on perceived acceptability of PWMI's participation in training and supervision, intervention fidelity and contagion, assessment of randomization, and feasibility and psychometric properties of outcome measures in a cluster design. Secondary objectives are change in provider and patient outcomes. The control condition is existing mental health training and supervision for non-specialists delivered through the Programme for Improving Mental Healthcare (PRIME), which includes the mental health Global Action Programme (mhGAP) and psychosocial treatments. The intervention condition will incorporate social contact with PWMI into existing PRIME training and supervision. Participants in the pilot will be the direct beneficiaries of training and supervision (i.e., primary care workers) and indirect beneficiaries (i.e., their patients). Primary care workers' outcomes include knowledge (mhGAP knowledge scale), explicit attitudes (mhGAP attitudes and social distance scales), implicit attitudes (Implicit Association Test), and clinical competence (Enhancing Assessment of Common Therapeutic factors, ENACT) to be assessed pre-training, post-training, and at 4-month follow-up. Patient outcomes include functioning, stigma experiences in accessing care, and depression/alcohol use symptoms to be assessed at initiation of mental health care and 6 months later. The pilot study will assist in modifying the intervention to inform a larger effectiveness trial of RESHAPE to ultimately improve provider attitudes and clinical competence as a mechanism to improve patient outcomes.

DETAILED DESCRIPTION:
Setting The study will take place in primary care health facilities in Chitwan, Nepal. The Department for International Development (DFID)-sponsored Programme for Improving Mental Health Care (PRIME) is being implemented in Chitwan, Nepal. PRIME aims to improve the coverage of treatment for priority mental disorders by implementing and evaluating a comprehensive mental health care package, integrated into primary health care in five low and middle income countries (LMIC) (Nepal, India, South Africa, Ethiopia and Uganda). The care package includes the provision of psychosocial and pharmacological interventions by non-specialized primary health workers (following the World Health Organization mental health Gap Action Programme (mhGAP)-Intervention Guide) and community counselors. Currently, no mental health services are systematically available in primary health care.

The facilities include health posts, primary health centers, and urban clinics. These are all part of the government health center and represent the first portal for care. In these facilities, primary care providers refer to health auxiliaries staff: health assistants, community medical assistants, and auxiliary nurse midwives. PRIME and the RESHAPE component are conducted by Transcultural Psychosocial Organization (TPO) Nepal, a Nepali non-governmental mental health research and training organization.

Design The investigator will use a pilot cluster randomized trial design. Because attitudes and clinical behaviors are influenced by peers (reference), the investigator anticipates a high degree of contagion among providers within a facility. Moreover, clinical care is not restricted to exclusive relationships with a single provider in the government health system. Therefore, patient care will be characterized by seeing a range of providers within a single facility over the course of their treatments. Therefore, a cluster design with the health facility as the unit of clustering is required.

Interventions The control arm will include the standard PRIME training and supervision protocol for Nepal. There are two versions of the PRIME training: one for prescribers and one for non-prescribers. Prescribers refer to health workers who can prescribe medication (health assistants and auxiliary health workers). Non-prescribers cannot prescribe medication and provide community outreach, assist in vaccination within maternal and child health programs, and promote adherence. Non-prescribers are predominantly auxiliary nurse midwives. Training for prescribers is based on mhGAP and includes target disorders of depression, psychosis, epilepsy, and harmful drinking. Psychosocial modules focusing on communication skills, supportive techniques, and health education are included based on prior curriculums and adapted for Nepal. Training is delivered by a psychiatrist and an experienced psychosocial counselor. Following training, the prescriber group participates in monthly supervision sessions with a psychiatrist. Non-prescribers receive training which includes psychosocial basics, a modified behavioral activation module, and a modified motivational interviewing module. These later psychological treatments, known as Healthy Activity Program (HAP) and Counseling for Alcohol Programs (CAP) respectively, have been developed for use in South Asia by non-specialists. Non-prescribers receive monthly supervision from experienced psychosocial counselors.

RESHAPE-mh uses the basic model of PRIME training and supervision. For both the prescriber and non-prescriber training, people with mental illness (PWMI) participate as co-facilitators. PWMI are trained to serve as co-facilitators using "PhotoVoice"-a participatory research approach in which photography is used to develop testimonials and other messaging. PWMI contribute to personal testimonials, ongoing social contact, myth busting, and provide a recovery emphasis. In addition, a health worker who has previously participated in the PRIME program receives training to participate as a co-facilitator and serves as an enthusiastic and aspirational role model. The second component of RESHAPE is ongoing engagement with PWMI through monthly consumer consultation meetings. [Note: In Duke Institutional Review Board (IRB) Pro00055042 and in National Institute of Mental Health (NIMH) grant application K01MH104310, RESHAPE is referred to as "Consumer Engagement Anti-Stigma (CEAS) Training." CEAS has now been renamed as RESHAPE-mh.]

Participants Primary care workers are the intended direct beneficiaries of RESHAPE. Their patients are the intended indirect beneficiaries. Primary care workers include prescribers (health assistants and auxiliary health workers) and non-prescribers (auxiliary nurse midwives) both of whom represent the first contact for most care needs. Medical doctors (MBBS) are limited to primary health centers and hospitals are usually seen after a person has encountered one of the lower level cadre of workers. In the pilot, additional participants will include PWMI who will be trained as facilitators for RESHAPE, mental health experts (psychiatrists and psychosocial counselors) who serve as facilitators and supervisors, and research staff (research assistants, field coordinators, and external competency and fidelity raters). For the pilot, the investigator plans to recruit all primary care workers (prescribers and non-prescribers) who are participating in the PRIME scale-up phase and a subset of their patients.

Randomization RESHAPE is a pilot cluster randomize trial. As mentioned, the reason for cluster randomization is because of the expected contagion at the level of the health facility. Health attitudes and behaviors are influenced by co-workers, and therefore the investigators expect that an intervention done with one health worker in a facility will influence peers. In addition, contagion may occur during other trainings among community health workers. Therefore, the health care provider randomization plan is to randomize all prescribers and non-prescribers associated with a specific facility.

Planned analyses

Qualitative analyses: Focus group discussions (FGD), cognitive interviews, and process evaluation notes will be coded in NVIVO (software name) and analyzed using content analysis for themes of cultural acceptability, experience of consumers as trainers, relevance to clinical care, training duration, structure of training, content of training, and follow-up engagement. Coding will be conducted among independent raters, and inter-rater reliability will calculated using Kappas. Data analysis will be conducted throughout each step to facilitate iterative revision then finalization of the manual.

Statistical analyses: The quantitative outcomes of interest will be summarized descriptively and visually over time for the providers (4 time points: pre- and post-training, then 4 months later, followed by another 12 months after that assessment point) and patients (2 time points: study entry and 6 months later) for both study arms. Total and validated domain-specific scores will be obtained for each instrument. Patient (PT)-specific trends over time for each score will be plotted to examine between-PT differences and to determine the plausible pattern (e.g. linearity) of those trends. This information will be used to inform the choice of effect estimate (e.g. difference in slopes or in means at a specific follow-up time point) in a subsequent cluster-randomized trial (C-RCT). The profiles will be grouped by cluster and by study arm to examine between-cluster and between-arm variation in PT outcomes. Using the first PT measurement (i.e. in the absence of intervention), preliminary estimates of within- and between-cluster variances, within- and between-primary care workers (PCW) variances and the intra-class correlation coefficient (ICC) of PT outcomes will be estimated. Such estimates are essential for sample size calculations for the planned R01 C-RCT design. Such variances are often guessed or obtained from other studies, whereas the investigator will obtain context and design-specific estimates using this pilot data. Moreover, the investigator will be able to estimate variance components for other measures of interest, such as PT-specific slopes, as appropriate. PCW-specific trends for each PCW-score will be examined using the same strategy as for PTs. Preliminary indicative estimates of differences in perceptions by arm will be obtained. Because the proposed K01 study is a pilot, no hypothesis-based inference testing will be performed. Instead, all quantitative analyses will focus on description. Analyses will be used for publication on the C-RCT pilot and for modification for full-scale C-RCT.

Ethics and research governance Consent: Providers will be told in the consent form that there are two different training approaches being evaluated. They will not be told about the focus regarding stigma as this may bias the outcomes. Nor will they be told that the main difference between trainings is the presence of PWMI as co-facilitators as this may contribute to attentional biases.

Harms: The main risk factor is psychological distress among consumers depending on the type of interaction with health care trainees in the training. If consumers do not feel that the engagement training is comfortable training environment, the investigator has outlined contingency plans regarding use of videotaped testimonials. Given a prior training with healthcare consumers in Nepal, the investigator anticipates that consumers will find the training experience a non-distressing experience. Minimal risk of harm from the treatment is anticipated. If patients require medication, hospitalization, or treatment, they will continue to be followed. Thus, there is not a disincentive for patients or providers to transition to other care if needed. In addition to these risks with greatest likelihood, other issues to consider are 1) negative consequences if confidentiality of information obtained in the study (including subject identity as a research participant or information collected during assessments or abstracted from a medical record review) were compromised.

Treatment for patients in the study is at the discretion of PCWs. PCW training includes both psychotherapy and medication management. At any time, PCWs may decide to initiate medication. All patients are expected to be receiving optimal clinical care at the clinical judgment of PCWs. PCWs are supervised by psychiatrists in Chitwan who can provide information on management and receive referrals for patients with worsening symptoms or other clinical concerns. All changes in treatment resulting from Adverse Events or Serious Adverse Events will be reported to institutional review boards.

Research ethics approval: This protocol has been approved by Duke University (Protocol Number: Pro00055042) and the Nepal Health Research Council (Regulatory Number: 110/2014).

Amendments: Amendments will be jointly reviewed by Duke University and Nepal Health Research Council, as well submitted to the funder: the National Institute of Mental Health, USA.

Timescale Trainings for PRIME and PRIME plus RESHAPE will take place in February-June 2016. Providers will be followed for two years to evaluate retention, changes in knowledge, attitudes, and clinical competence. Patient will be enrolled at facilities approximately 18 months after training. They will be followed-up six months after initial enrollment evaluation. Primary outcome data collection will be completed by the end of June 2018.

ELIGIBILITY:
Participant Types

* Primary care workers (primary beneficiary)
* Patients (indirect beneficiary)

Inclusion Criteria:

* All primary care workers participating in either the prescriber or non-prescriber PRIME trainings will be invited to participate
* Primary care trainees will need to be 21-65 years of age
* Recruitment will attempt to balance gender distribution in the recruitment health clusters
* All participants will need to have Nepali language competency, be actively engaged in care provision in their health cluster, and have a valid certificate of practice from the Ministry of Health
* Primary care trainees need to have permission from their health supervisor to attend the entire duration of the training.
* Any patient receiving PRIME services will be invited to participate. This includes persons with diagnoses of depression, psychosis, harmful drinking, or epilepsy. Providers make the diagnosis based on mhGAP criteria.
* For patients, inclusion criteria will be 21-65 years of age and fluency in Nepali.

Exclusion Criteria:

* Primary care trainees will be excluded if they have any prior citations on their clinical practice licensure.
* Patients who cannot provide consent will be excluded.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in stigmatizing attitudes, as measured by the Social Distance questionnaire | Baseline, post-training (immediately after 10-day training curriculum), +4 months, + 16 months
  Health Provider Outcome: Health providers rate the degree of social distance from persons with mental illness related to 10 domains, e.g., willingness to work together, willingness to be friends, willingness to share meals

SECONDARY OUTCOMES:
Change in clinical knowledge, as measured by the mhGAP knowledge assessment | Baseline, post-training (immediately after 10-day training curriculum), +4 months, + 16 months
  Health Provider Outcome: Clinical knowledge is assessed with the mhGAP knowledge assessment multiple choice evaluation.
Change in patient functioning, as measured by the World Health Organization Disability Assessment Scale (WHODAS) | Baseline, 6 months
  Patient Outcome: Patient functioning is assessed with the World Health Organization Disability Assessment Scale (WHODAS). This is the primary measure of interest for patient outcomes.
Change in patient perceived stigma as a barrier to accessing care, as measured by the Barriers to Access to Care Evaluation (BACE) | Baseline, 6 months
  Patient Outcome: Patient perceived stigma is assessed with the Barriers to Access to Care Evaluation (BACE)
Change in implicit attitudes, as measured by the Implicit Association Test (IAT) | Baseline, +4 months, + 16 months
  Health Provider Outcome: Implicit Association Test (IAT) of implicit biases associating mental disorders versus physical disorders on attributes of harmfulness vs. harmlessness
Change in patient depression, as measured by the Patient Health Questionnaire (PHQ-9) | Baseline, 6 months
  Patient Outcome: Clinically and culturally validated version of the PHQ-9 to measure depression symptom severity
Change in stigmatizing attitudes, as measured by the mhGAP Attitudes Questionnaire | Baseline, post-training (immediately after 10-day training curriculum), +4 months, + 16 months
  Health Provider Outcome: attitudinal questions related to mental illnesses including depression, psychosis, epilepsy, and alcohol use
Change in clinical competence, as measured by Enhancing Assessment of Common Therapeutic factors | Baseline, +4 months, + 16 months
  Health Provider Outcome: Clinical competence is assessed with the Enhancing Assessment of Common Therapeutic factors. The ENACT is scored through observed or recorded role plays between primary care workers and standardized patients.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon A Kohrt, MD, PhD, Principal Investigator — George Washington University
Locations (1):
- Transcultural Psychosocial Organization (TPO) Nepal, Bharatpur, Chitwan, Nepal

REFERENCES:
- [Background] Kohrt BA, Luitel NP, Acharya P, Jordans MJ. Detection of depression in low resource settings: validation of the Patient Health Questionnaire (PHQ-9) and cultural concepts of distress in Nepal. BMC Psychiatry. 2016 Mar 8;16:58. doi: 10.1186/s12888-016-0768-y. PMID 26951403
- [Background] Jordans MJ, Kohrt BA, Luitel NP, Komproe IH, Lund C. Accuracy of proactive case finding for mental disorders by community informants in Nepal. Br J Psychiatry. 2015 Dec;207(6):501-6. doi: 10.1192/bjp.bp.113.141077. Epub 2015 Oct 8. PMID 26450582
- [Background] Griffith JL, Kohrt BA. Managing Stigma Effectively: What Social Psychology and Social Neuroscience Can Teach Us. Acad Psychiatry. 2016 Apr;40(2):339-47. doi: 10.1007/s40596-015-0391-0. Epub 2015 Jul 11. PMID 26162463
- [Background] Kohrt BA, Jordans MJ, Rai S, Shrestha P, Luitel NP, Ramaiya MK, Singla DR, Patel V. Therapist competence in global mental health: Development of the ENhancing Assessment of Common Therapeutic factors (ENACT) rating scale. Behav Res Ther. 2015 Jun;69:11-21. doi: 10.1016/j.brat.2015.03.009. Epub 2015 Mar 24. PMID 25847276
- [Background] Kohrt BA, Hruschka DJ. Nepali concepts of psychological trauma: the role of idioms of distress, ethnopsychology and ethnophysiology in alleviating suffering and preventing stigma. Cult Med Psychiatry. 2010 Jun;34(2):322-52. doi: 10.1007/s11013-010-9170-2. PMID 20309724
- [Background] Kohrt BA, Tol WA, Harper I. Reconsidering somatic presentation of generalized anxiety disorder in Nepal. J Nerv Ment Dis. 2007 Jun;195(6):544; author reply 545. doi: 10.1097/NMD.0b013e318064e7eb. No abstract available. PMID 17568305
- [Background] Kohrt BA, Harper I. Navigating diagnoses: understanding mind-body relations, mental health, and stigma in Nepal. Cult Med Psychiatry. 2008 Dec;32(4):462-91. doi: 10.1007/s11013-008-9110-6. PMID 18784989
- [Background] Jordans MJ, Luitel NP, Pokhrel P, Patel V. Development and pilot testing of a mental healthcare plan in Nepal. Br J Psychiatry. 2016 Jan;208 Suppl 56(Suppl 56):s21-8. doi: 10.1192/bjp.bp.114.153718. Epub 2015 Oct 7. PMID 26447173
- [Background] Makan A, Fekadu A, Murhar V, Luitel N, Kathree T, Ssebunya J, Lund C. Stakeholder analysis of the Programme for Improving Mental health carE (PRIME): baseline findings. Int J Ment Health Syst. 2015 Jul 8;9:27. doi: 10.1186/s13033-015-0020-z. eCollection 2015. PMID 26155307
- [Background] Luitel NP, Jordans MJ, Adhikari A, Upadhaya N, Hanlon C, Lund C, Komproe IH. Mental health care in Nepal: current situation and challenges for development of a district mental health care plan. Confl Health. 2015 Feb 6;9:3. doi: 10.1186/s13031-014-0030-5. eCollection 2015. PMID 25694792
- [Background] Brenman NF, Luitel NP, Mall S, Jordans MJ. Demand and access to mental health services: a qualitative formative study in Nepal. BMC Int Health Hum Rights. 2014 Aug 2;14:22. doi: 10.1186/1472-698X-14-22. PMID 25084826
- [Derived] Kaiser BN, Gurung D, Rai S, Bhardwaj A, Dhakal M, Cafaro CL, Sikkema KJ, Lund C, Patel V, Jordans MJD, Luitel NP, Kohrt BA. Mechanisms of action for stigma reduction among primary care providers following social contact with service users and aspirational figures in Nepal: an explanatory qualitative design. Int J Ment Health Syst. 2022 Aug 11;16(1):37. doi: 10.1186/s13033-022-00546-7. PMID 35953839
- [Derived] Kohrt BA, Jordans MJD, Turner EL, Rai S, Gurung D, Dhakal M, Bhardwaj A, Lamichhane J, Singla DR, Lund C, Patel V, Luitel NP, Sikkema KJ. Collaboration With People With Lived Experience of Mental Illness to Reduce Stigma and Improve Primary Care Services: A Pilot Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2131475. doi: 10.1001/jamanetworkopen.2021.31475. PMID 34730821
- [Derived] Rai S, Gurung D, Kaiser BN, Sikkema KJ, Dhakal M, Bhardwaj A, Tergesen C, Kohrt BA. A service user co-facilitated intervention to reduce mental illness stigma among primary healthcare workers: Utilizing perspectives of family members and caregivers. Fam Syst Health. 2018 Jun;36(2):198-209. doi: 10.1037/fsh0000338. PMID 29902036
- [Derived] Kohrt BA, Jordans MJD, Turner EL, Sikkema KJ, Luitel NP, Rai S, Singla DR, Lamichhane J, Lund C, Patel V. Reducing stigma among healthcare providers to improve mental health services (RESHAPE): protocol for a pilot cluster randomized controlled trial of a stigma reduction intervention for training primary healthcare workers in Nepal. Pilot Feasibility Stud. 2018 Jan 24;4:36. doi: 10.1186/s40814-018-0234-3. eCollection 2018. PMID 29403650

DOCUMENTS (1):
  • Informed Consent Form (2014-05-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02793271/ICF_000.pdf